CLINICAL TRIAL: NCT03710174
Title: Evaluation of the Effectiveness of Infrared LED Photobiomodulation in Children With Sleep Bruxism: Study Protocol for Randomized Clinical Trial.
Brief Title: Evaluation of the Effectiveness of Infrared LED Photobiomodulation in Children With Sleep Bruxism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fernanda Yukie Kobayashi, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ferbruxismo
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Bruxism, Sleep
MeSH Terms: conditions — Sleep Bruxism | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not know to which group the participants belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Without bruxism and no intervention. They will be submitted to electromyographic assessment and evaluation of salivary cortisol and dopamine.
- LED group (Experimental): The volunteers in Group 2 will be submitted to the initial evaluation of the morphological and psychosocial variables. During the same appointment, red LED (3 X 6 cm) will be administered using a board with 6 LEDs with a wavelength of 650 nm ± 20 nm, seven-minute operation time, optical spot of 5 ± 2 mm and optical output of 2~5 mW, with a dose of 2.675 J/cm2. Further analyses will be performed immediately after the photobiomodulation session and one week later. They will be submitted before and after LED to electromyographic assessment and evaluation of salivary cortisol and dopamine.
  Interventions: Radiation: Infrared LED photobiomodulation
- Occlusal splint group (Experimental): They will be treated using the standard protocol of a rigid occlusal splint. After the initial evaluation, molds will be made for the fabrication of the splints, which will be delivered one week later. Written and verbal instructions for use will be given. After one month of daily use, the volunteers will return for the final morphological and psychosocial evaluations.
  Interventions: Device: Occlusal splint
- Placebo group (Placebo Comparator): Subjects with bruxism. The same procedures as LED group, but the device will be turn off.
  Interventions: Radiation: Placebo LED photobiomodulation

INTERVENTIONS:
Radiation: Infrared LED photobiomodulation — Infrared LED (3 X 6 cm) will be administered using a board with 6 LEDs with a wavelength of wavelength: 850 nm ± 20 nm, seven-minute operation time, optical spot of 5 ± 2 mm and optical output of 2~5 mW, with a dose of 2.675 J/cm2. Further analyses will be performed immediately after the photobiomodulation session and one week later.
  Arms: LED group
Device: Occlusal splint — After the initial evaluation, molds will be made for the fabrication of the splints, which will be delivered one week later. Written and verbal instructions for use will be given. After one month of daily use, the volunteers will return for the final morphological and psychosocial evaluations.
  Arms: Occlusal splint group
Radiation: Placebo LED photobiomodulation — The same procedure as LED group with the device turned off.
  Arms: Placebo group

SUMMARY:
Sleep bruxism is a masticatory muscle activity characterized as rhythmic (phasic) or non-rhythmic (tonic). The literature reports the prevalence rates, diverse etiologies and different types of treatment. In children and adolescents, etiological factors, such as breathing pattern and sleep quality, have recently been addressed in studies investigating sleep bruxism. While studies have also reported psychological factors as a causal factor, this aspect requires further research. There are also divergences in opinion regarding the form of treatment. New therapies for adults, such as botulinum toxin, have been investigated, but such techniques are not applicable for individuals in the growth and development phase. Thus, photobiomodulation therapy has piqued the interest of researchers, as this noninvasive method has demonstrated positive results in problems related to muscle tissues. This document describes the protocol for a proposed study to evaluate morphological and psychosocial aspects in children and adolescents with awake bruxism and their responses to photobiomodulation therapy with infrared LED.

ELIGIBILITY:
Inclusion Criteria:

* mixed dentition phase (permanent incisors and molars erupted)
* established permanent dentition.

Exclusion Criteria:

* dental caries
* using medications, such as anti-inflammatory agents, muscle relaxants, corticoids, anticonvulsants and antidepressants
* those with chronic diseases that affect muscles or motor coordination
* those who do not cooperate during the evaluation

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in muscle activity evaluated by electromyography | Before and immediately after treatment
  Electromyography will be performed to complement the evaluation of the morphological aspects of the groups. The masseter and temporal muscles will be evaluated using a portable electromyograph (BTS TMJOINT) with wireless electrodes. The participant will be seated with Camper's plane parallel to the floor. Three readings will be made on both sides with the muscles at rest, during habitual maximum intercuspation (isometric contraction) and during simulated chewing with Parafilm (isotonic contraction). The signal will be captured for 10 seconds under each condition. The first chewing cycle will be discarded and the subsequent five cycles will be collected.

SECONDARY OUTCOMES:
Change in salivary cortisol and dopamine | Before and immediately after treatment
  The participants and caregivers will receive verbal and written instructions to avoid any physical activity, the ingestion of substances with alcohol or caffeine, soft drinks, tea, corticoids and chewing gum in the 24h prior to the collection of the saliva. Saliva samples will be collected using swabs, which will refrigerated immediately after collection. The swab will be placed under the tongue. Samples with visible signs of blood will be discarded due to possible contamination. The swabs will be centrifuged at 3500 rpm for 5 minutes. The supernatant will be collected and stored at -40o C. Cortisol will be determined using an enzyme-linked immunosorbent assay. Dopamine will also be determined using an ELIZA kit. The samples will be thawed and centrifuged again. The procedure will follow the basic ELISA principle of competition between an untagged antigen and an enzyme-tagged antigen for a particular number of binding sites on the antibody.

CONTACTS AND LOCATIONS:
Locations (1):
- Uninove, São Paulo, São Paulo, Brazil